CLINICAL TRIAL: NCT02926222
Title: Regorafenib in Relapsed Glioblastoma REGOMA Study Randomized, Controlled Open-label Phase II Clinical Trial
Brief Title: Regorafenib in Relapsed Glioblastoma
Acronym: REGOMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: BAYER S.p.A. - Italia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-GB-1-2014 REGOMA; 2014-003722-41 (EudraCT Number)
Record Dates: First submitted 2016-06-22; First posted 2016-10-06 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — regorafenib; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A - Regorafenib (Experimental): Patients receive REGORAFENIB 40 mg tablets once daily (160 mg/die), 3 weeks on, 1 week off, until disease progression or unacceptable toxicity.
  Interventions: Drug: Regorafenib
- ARM B - Lomustine (Active Comparator): Patients receive LOMUSTINE 110 mg/m2 orally on day 1, every 6 weeks (q6w), until disease progression or unacceptable toxicity.
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: Regorafenib — Regorafenib is formulated as tablets of 40mg for oral administration.
  Other Names: Stivarga
  Arms: ARM A - Regorafenib
Drug: Lomustine — Lomustine is formulated as tablets of 40mg for oral administration.
  Other Names: Ceenu
  Arms: ARM B - Lomustine

SUMMARY:
This study aims to evaluate the role of Regorafenib in prolonging the overall survival of glioblastoma multiforme patients who progressed after surgery and Stupp regimen with or without bevacizumab.

DETAILED DESCRIPTION:
The primary aim of the study is to evaluate the overall survival (OS) in the intention to treat (ITT) population. Secondary aims are to evaluate the progression free survival (PFS), safety, objective response rate (ORR), disease control rate (DCR) in the ITT population, and the evaluation of quality of life (QoL). Additional exploratory objectives include the analysis of antiangiogenic and metabolic biomarkers in tissue at first and second surgery (if performed) by the evaluation of certain metabolic features of tumors that could be involved in tumor responses to antiangiogenic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Histologically confirmed de novo glioblastoma multiforme (grade IV)
* First recurrence after adjuvant treatment (surgery followed by radiotherapy and temozolomide chemotherapy with or without bevacizumab) in patients who have not received further therapeutic interventions
* For patients not undergoing a second surgery at the time of relapse, recurrent disease must include at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm, visible on 2 or more axial slices 5 mm apart, based on an MRI scan done within 2 weeks prior to randomization
* Documented progression of disease as defined by RANO criteria at least 12 weeks after completion of radiotherapy, unless the recurrence is outside the radiation field or has been histologically documented
* Have adequate bone marrow function, liver function, and renal function, as measured by the following laboratory assessments conducted within 7 days prior to the initiation of study treatment:

  * Hemoglobin >9.0 g/dl
  * Absolute neutrophil count (ANC) >1500/mm3 without transfusions or granulocyte colony stimulating factor and other hematopoietic growth factors
  * Platelet count ≥100,000/μl
  * White blood cell count (WBC) >3.0 x 109/L
  * Total bilirubin <1.5 times the upper limit of normal
  * ALT and AST <3 x upper limit of normal (<5 x upper limit of normal for patients with liver involvement of their cancer and/or have bone metastasis)
  * Serum creatinine <1.5 x upper limit of normal
  * Alkaline phosphatase <2.5 x ULN (<5 x upper limit of normal for patients with liver involvement of their cancer and/or have bone metastasis)
  * PT-INR/PTT <1.5 x upper limit of normal (Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists per medical history)
  * Lipase ≤ 1.5 x the ULN
* Glomerular filtration rate ≥ 30 mL/min/1.73 m2 according to the Modified Diet in Renal Disease abbreviated formula
* Analyses of MGMT methylation status on tumoral tissue at first surgery (at own institution)
* Understand, be willing to give consent, and sign the written informed consent form (ICF) prior to undergoing any study-specific procedure
* If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment
* If female and of childbearing potential, or if male, agree to use adequate contraception (eg, intrauterine device, oral contraceptive, or double-barrier method) based on the judgment of the investigator or a designated associate from the date on which the ICF is signed until 8 weeks after the last dose of study drug
* World Health Organization (WHO) Performance status ≤ 1 (or Karnofsky performance status (KPS) ≥70)) within 14 days prior to the initiation of study treatment
* Stable or decreasing dosage of steroids for 7 days prior to the baseline MRI scan.
* Patients may have undergone surgery for the recurrence; the histological report must document a glioblastoma recurrence. If operated:

  * at least 28 days and maximum 42 days interval from the surgery is required prior to administration of study drugs and patients should have fully recovered
  * Exclusion Criteria:
* Are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort)
* Radiotherapy within 12 weeks prior to the diagnosis of progression, if the lesion is in the radiation field,
* Have had systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and/or hormonal therapy within 4 weeks prior to initiation of study treatment
* Positioning of carmustin wafers during first or second surgery
* Other active or inactive malignancy (except for carcinoma in situ of the cervix, of the prostate or basal cell carcinoma). Malignancy will be considered inactive if patients are in complete remission for at least 3 years prior to study entry
* Have had prior treatment with regorafenib or any other VEGFR-targeting kinase inhibitor
* Have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment
* Are pregnant
* Are breastfeeding
* Are unable to swallow oral tablets (crushing of study treatment tablets is not allowed)
* Have congestive heart failure classified as New York Heart Association Class 2 or higher
* Have had unstable angina (angina symptoms at rest) or new-onset angina ≤ 3 months prior to screening.
* Have had a myocardial infarction < 6 months prior to initiation of study treatment
* Have cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin
* Have uncontrolled hypertension (systolic blood pressure [SBP] > 140 mmHg or diastolic blood pressure [DBP] > 90 mmHg) despite optimal medical management
* Have had arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within 6 months prior to the initiation of study treatment
* Have an ongoing infection with severity of Grade 2 or above (NCI-CTCAE v 4.0)
* Have a known history of human immunodeficiency virus infection
* Have either active or chronic hepatitis B or C requiring treatment with antiviral therapy
* Have a history of organ allograft
* Have evidence or history of any bleeding diathesis (including mild hemophilia), irrespective of severity
* Have had a hemorrhage or a bleeding event ≥ Grade 3 (NCI-CTCAE v 4.0) within 4 weeks prior to the initiation of study treatment
* Have a non-healing wound, ulcer, or bone fracture
* Have renal failure requiring hemodialysis or peritoneal dialysis
* Have dehydration ≥ Grade 1 (NCI-CTCAE v 4.0)
* Have interstitial lung disease with ongoing signs and symptoms at the time informed consent is obtained
* Have persistent proteinuria > 3.5 g/24 hours measured by urine protein creatinine ratio from a random urine sample (Grade 3, NCI-CTCAE v 4.0)
* Have any other serious or unstable illness, or medical, psychological, or social condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results
* Have a known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
* Have any malabsorption condition
* Recurrent disease located outside of the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to 18 months or to the date of death from any cause

SECONDARY OUTCOMES:
Progression free survival | From the date of randomization to 18 months or to the date of disease progression or to the date of death, whichever occurs first
Objective response rate | Approximately 36 months
  As percentage of patients achieving a complete response plus partial response
Disease control rate | Approximately 36 months
  As percentage of patients achieving a complete response plus partial response plus stable disease
Toxicity (Graded according to the NCI-Common Terminology Criteria for Adverse Events) | Approximately every 4 weeks through the treatment period up to 30 days after the end of treatment
  Graded according to the NCI-Common Terminology Criteria for Adverse Events (CTCAE) v.4

OTHER OUTCOMES:
Quality of life EORTC | From the date of randomization, approximately every 3 months until the date of first documented progression or date of death from any cause, or study withdrawal, whichever came first, assessed up to 30 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorina Zagonel, MD, Principal Investigator — Istituto Oncologico Veneto IRCCS
Locations (10):
- Italy (10):
  - IRCCS "Saverio de Bellis, Castellana Grotte, BA
  - Ospedale di Bellaria, Bologna, BO
  - Azienda Ospedaliera "G.Rummo", Benevento, BR
  - istituto Scientifico Romagnolo per lo Studio e Cura dei Tumori, Cesena, FC
  - Istituto Neurologico C. Besta IRCCS, Milan, MI
  - Istituto Oncologico Veneto IRCCS, Oncologia Medica 1, Padua, PD
  - Ospedale Santa Chiara, Pisa, PI
  - Azienda Ospedaliero Universitaria S. Maria della Misericordia, Udine, UD
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lombardi G, Del Bianco P, Brandes AA, Eoli M, Ruda R, Ibrahim T, Lolli I, Rizzato S, Daniele B, Pace A, Pasqualetti F, Caccesse M, Bergo E, Magni G, De Salvo GL, Zagonel V. Patient-reported outcomes in a phase II randomised study of regorafenib compared with lomustine in patients with relapsed glioblastoma (the REGOMA trial). Eur J Cancer. 2021 Sep;155:179-190. doi: 10.1016/j.ejca.2021.06.055. Epub 2021 Aug 10. PMID 34388515
- [Derived] Lombardi G, De Salvo GL, Brandes AA, Eoli M, Ruda R, Faedi M, Lolli I, Pace A, Daniele B, Pasqualetti F, Rizzato S, Bellu L, Pambuku A, Farina M, Magni G, Indraccolo S, Gardiman MP, Soffietti R, Zagonel V. Regorafenib compared with lomustine in patients with relapsed glioblastoma (REGOMA): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2019 Jan;20(1):110-119. doi: 10.1016/S1470-2045(18)30675-2. Epub 2018 Dec 3. PMID 30522967